CLINICAL TRIAL: NCT07127224
Title: Consciousness Prognosis Evaluation Using Olfactory Stimulations in Comatose Patients
Brief Title: Consciousness Prognosis Evaluation Using Olfactory Stimulations in Comatose Patients)
Acronym: CEOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: D21-P017
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Disorders of Consciousness Due to Severe Brain Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with disorders of consciousness (Experimental): Adult ICU patients with disorders of consciousness will undergo non-invasive neurophysiological assessments including olfactory, auditory, and somatosensory stimulations. Olfactory stimuli are added for prognostic evaluation. Clinical and neurological follow-up will be done at 3 months.
  Interventions: Diagnostic Test: Olfactory stimulation

INTERVENTIONS:
Diagnostic Test: Olfactory stimulation — Olfactory stimulation ("sniff" test) combined with auditory and somatosensory stimulations during bedside neurophysiological assessments to evaluate neurological prognosis in ICU patients.

SUMMARY:
The goal of this observational study is to determine whether the clinical response to olfactory stimulation (known as the "sniff" response) can help predict 3-month neurological outcomes in ICU patients with persistent disorders of consciousness after sedation withdrawal, regardless of the reason for admission or the initial severity.

The main questions this study aims to answer are:

* Can the "sniff" response to olfactory stimulation predict neurological outcomes at 3 months?
* Is this response a better prognostic indicator than commonly used neurophysiological tests? Researchers will compare the results obtained from olfactory stimulation with those from somatosensory and auditory stimulations to determine whether the olfactory method provides additional or superior prognostic value.

Participants will receive additional olfactory stimuli as part of the neurophysiological evaluation for prognostic purposes and be followed up at 3 months for clinical, neurological, and functional evaluation

ELIGIBILITY:
Inclusion Criteria:

* Admission to neuro-intensive care unit (neuro-ICU)
* Age ≥ 18 years
* Patients with persistent disorders of consciousness defined by an abnormal CRS-R score (<16) at 72 hours after sedation withdrawal and spontaneous ventilation
* Consent obtained from legal representatives or activation of emergency waiver
* Patient covered by or affiliated with a social security system

Exclusion Criteria:

* Pregnancy
* Brain death
* Pre-existing ENT or olfactory bulb pathologies that may affect olfactory functions
* Acute or chronic peripheral neurological diseases that may alter evoked potentials
* Known neurodegenerative diseases (e.g., Parkinson's disease, Alzheimer's disease)
* Patients under legal guardianship or protective supervision (safeguard or protection measures)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2027-05-05 (Estimated); Study Completion 2027-05-05 (Estimated)

PRIMARY OUTCOMES:
Glasgow Outcome Scale-Extended (GOS-E) score at 3 months | 3 months after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- GHU Psychiatrie et Neurosciences, Paris, GHU Psychiatrie Et Neurosciences, France

IPD SHARING:
Plan to Share IPD: Undecided